CLINICAL TRIAL: NCT03187236
Title: The Early Detection, Clinical Course and Prognosis of Anxiety and Depression in Chronic Obstructive Pulmonary Disease
Brief Title: Registry for Chronic Obstructive Pulmonary Disease With Anxiety and Depression in China
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Jianguo He, Chief of Pulmonary Vascular Disease Center, Chinese Academy of Medical Sciences, Fuwai Hospital
Other Study IDs: 2016YFC1304404A
Record Dates: First submitted 2017-06-13; First posted 2017-06-14 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: COPD; Anxiety; Depression
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Anxiety Disorders; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Serum and blood cells
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Anxiety and depression are common comorbidities of chronic obstructive pulmonary disease (COPD). However, the exact prevalence is not known in China. COPD patients with anxiety and depression tend to have more severe symptoms and worse prognosis, but the related evidences are not strong enough. The study aim to investigate the prevalence and long-term outcome of anxiety and depression in COPD.

ELIGIBILITY:
Inclusion Criteria:

* Stable chronic obstructive pulmonary disease (COPD) patients

Exclusion Criteria:

* Patients with bronchial asthma or other severe pulmonary diseases or having received pulmonary surgery in 6 months
* Patients with tumor history during past 5 years
* Patients with COPD exacerbations during past 4 weeks
* Participants in clinical trials
* Patients in pregnancy or breastfeeding
* Patients unable to complete questionaire independently
* Patients older than 80 years old
* Patients receiving long-term domiciliary oxygen therapy

Max Age: 80 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Stable COPD patients
Sampling Method: Non-Probability Sample
Enrollment: 1906 (Estimated)
Dates: Start 2017-06-15 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
moderate and severe COPD exacerbations | 3 years
  total times

SECONDARY OUTCOMES:
All-cause mortality | 3 years
  mortality in %

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zhao X, Su R, Hu R, Chen Y, Xu X, Yuan Y, Zhang J, Zhang W, Yang Y, Chen M, Li D, Wu B, Huang D, Wu D. Sarcopenia index as a predictor of clinical outcomes among older adult patients with acute exacerbation of chronic obstructive pulmonary disease: a cross-sectional study. BMC Geriatr. 2023 Feb 11;23(1):89. doi: 10.1186/s12877-023-03784-7. PMID 36774462